CLINICAL TRIAL: NCT01305187
Title: Monocentric, Randomized, Subject and Rater Blinded Clinical Investigation to Prove the Non-inferiority of Belotero® Basic Versus Juvéderm® Ultra 3 Containing Lidocaine - After Single Injection for Correction of Nasolabial Folds (NLF)
Brief Title: Non-inferiority of Belotero® Basic Versus Juvéderm® Ultra 3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Dr. Matthias Zerm, Manager Public Disclosure, Merz Pharmaceuticals GmbH
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 90028_4007_0
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Physiological Stress; Disorder of Aging; Skin Diseases; Wrinkles; Nasolabial Folds
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyaluronic Acid Filler - Medical Device (Experimental)
  Interventions: Device: Hyaluronic Acid Filler

INTERVENTIONS:
Device: Hyaluronic Acid Filler — The dosage is individualized depending on the depth of the NLF. The goal is to achieve optimal correction of both NLF with single implantations of Belotero® Basic and Juvéderm® Ultra 3 respectively. Each subject will be injected with Belotero® Basic and Lidocaine containing Juvéderm® Ultra 3 according to a split-face design. The allocation of fillers to the side of the face will be randomized. The randomization method is block-wise with a ratio 1:1 to the groups Belotero® Basic left and Juvéderm® Ultra 3 right, Belotero® Basic right and Juvéderm® Ultra 3 left.

SUMMARY:
This study will investigate the non-inferiority of Belotero® Basic versus Juvéderm® Ultra 3 in the treatment of nasolabial folds

ELIGIBILITY:
Inclusion Criteria:

* Subject with bilateral, symmetrical NLF and wish for correction. Documented severity of NLF score 2 or 3 at screening on the Merz Wrinkle Severity Rating Scale II

Exclusion Criteria:

* Any severe or uncontrolled systemic disease (e.g. cardiac, renal, pulmonary, hepatic, or gastrointestinal). Subject suffering from diabetes mellitus, autoimmune and rheumatic diseases, clinically relevant coagulation disorders, recurrent angina, or severe psychic, neurological or mental disease
* History of malignancy within the last 5 years before the study
* Infection, inflammations or active dermatological disease in the face

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects reporting an equal or better outcome for the side of face treated with Belotero® Basic compared to the side of face treated with Juvéderm® Ultra 3 at V4 on the validated Wrinkle Severity Rating Scale II | Week 4

SECONDARY OUTCOMES:
Overall intra-individual change at V2 post implantation in the validated Wrinkle Severity Rating Scale II compared to V2 pre implantation | Week 0
Overall intra-individual change at V3 post implantation in the validated Wrinkle Severity Rating Scale II compared to V2 pre implantation | 2 Weeks
Overall intra-individual change at V4 post implantation in the validated Wrinkle Severity Rating Scale II compared to V2 pre implantation | 4 Weeks
Overall absolute score change at V2 post implantation in the validated Wrinkle Severity Rating Scale II compared to V2 pre implantation assessed by photo rating of one independent rater | Week 0
Overall absolute score change at V3 post implantation in the validated Wrinkle Severity Rating Scale II compared to V2 pre implantation assessed by photo rating of one independent rater | 2 Weeks
Overall absolute score change at V4 post implantation in the validated Wrinkle Severity Rating Scale II compared to V2 pre implantation assessed by photo rating of one independent rater | 4 Weeks
Proportion of overall responders i.e. at least 1 point improvement in the validated Wrinkle Severity Rating Scale II(WSRS II) at V4, based on the intra-individual change in WSRS II compared to baseline before implantation, V2 pre implantation | 4 Weeks
Assessment of Global aesthetic improvement [GAIS] by the investigator and subject V2 post implantation and V4 | 4 Weeks
Overall GAIS by photo rating of an individual rater V2 post implantation and V4 | 4 Weeks
Subject Satisfaction Questionnaire results at V2 pre and post implantation | Week 0
Subject Satisfaction Questionnaire results at V3 | 2 Weeks
Subject Satisfaction Questionnaire results at V4 | 4 Weeks
Global assessment of subject comfort at V2 post implantation by the investigator and the subject. | Week 0
Global assessment of subject comfort at V3 by the investigator and the subject | 2 Weeks
Global assessment of subject comfort at V4 by the investigator and the subject | 4 Weeks
Proportion of subjects feeling the implant at V2 post implantation | Week 0
Proportion of subjects feeling the implant at V3. | 2 Weeks
Proportion of subjects feeling the implant at V4 | 4 Weeks
Proportion of subjects recommending Belotero® Basic only or Juvéderm® Ultra 3 only or both at V4 | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Acker, Dr., Study Director — Merz Pharmaceuticals GmbH
Locations (1):
- Praxisklinik Kaiserplatz, Frankfurt am Main, Germany